CLINICAL TRIAL: NCT07096700
Title: Virtual Reality for Gait Training in Multiple Sclerosis (VIRTUE): an Interventional Feasibility Study
Brief Title: VR and Orthoses for Rehabilitation in Multiple Sclerosis
Acronym: VIRTUE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: VIRTUE
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Neurorehabilitation; Gait impairments; Virtual Reality; Wearable technology; Sensor-based monitoring; Inertial sensors; Physiological signals; Walking braces; Remote monitoring
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR - Multiple Sclerosis (Other): Twelve adults with multiple sclerosis who require a walking brace to support ambulation and are compatible with Virtual Reality
  Interventions: Other: VR and walking brace-based gait rehabilitation

INTERVENTIONS:
Other: VR and walking brace-based gait rehabilitation — The study implements the use of VR and wearable sensors to enhance gait analysis in clinical practice. Participants will take part in two outpatient sessions (T1 and T2) involving the use of VR and wearable sensors, during which they will be asked to complete standardized gait tests and questionnaires. These two sessions will be separated by a one-week home phase (Th), during which participants will wear the walking brace in their daily activities and their gait and physiological data will be recorded by wearable sensors. A final session (T3), conducted without VR, will be scheduled two months later to assess the long-term retention of the intervention effects.

SUMMARY:
This non-drug, non-medical device, interventional study explores the feasibility of integrating virtual reality (VR) with wearable sensors to support gait training using a passive orthosis in individuals with multiple sclerosis (MS). The aim is to determine whether this approach can enhance clinical gait assessment and facilitate orthosis adaptation by replicating real-life scenarios within a safe and controlled environment. The virtual environment, accessed through a head-mounted display, will be delivered via a custom simulator incorporating standardized gait tasks embedded in everyday settings. This system is designed to minimize the artificial influence of clinical settings on walking performance, while providing clinicians with objective gait data for more comprehensive evaluation.

DETAILED DESCRIPTION:
Patients with multiple sclerosis (MS) often experience significant gait impairments that impact their autonomy and overall quality of life. One of the primary rehabilitation strategies involves the use of walking braces. While these orthotic devices can support ambulation, their effective integration into daily life typically requires a period of adaptation and specific training. Traditionally, gait training and orthosis prescription occur in clinical settings, which may not fully reflect the real-world challenges that patients encounter. Moreover, current clinical assessments rely primarily on subjective observations and standardized scales, which may lack the sensitivity and objectivity needed to capture the full complexity of gait performance.

virtual reality (VR) offers a promising opportunity to simulate realistic walking environments in a controlled and safe setting, such as an outpatient clinic, potentially enhancing the outcomes of gait rehabilitation. Another promising technology in this domain is the use of wearable inertial sensors, which have been shown to effectively measure gait and postural parameters in people with MS. A further challenge associated with the use of orthotic devices is the physical and psychological stress they may cause, which can lead patients to discontinue their use. To evaluate such discomfort more objectively, recent studies have explored the use of physiological signal analysis and machine learning (ML) algorithms as an alternative or complement to self-reported questionnaires.

The integration of VR with wearable inertial and physiological sensors may allow for a more comprehensive and objective assessment of a patient's adaptation to walking braces. However, no validated system currently exists that combines these technologies for gait assessment and training with passive orthoses in people with MS.

The VIRTUE study aims to address this gap by developing and evaluating a VR-based platform (VIRTUE4MS) that replicates real-life scenarios, such as navigating through a museum, park, or grocery store, and enables standardized gait assessments within immersive environments. The system will employ both inertial and physiological wearable sensors to gather data on gait dynamics and user experience, ultimately supporting clinical decision-making regarding orthotic use. In this study, 12 patients with MS will perform walking and balance tasks over three sessions (T1, T2, T3), both with and without the Exoband brace, in VR and real-world conditions. Ultimately, this study seeks to explore an innovative, technology-supported approach to orthosis assessment and gait training that could complement traditional clinical tools and contribute to more effective, personalized rehabilitation strategies for individuals with MS.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple sclerosis
* Age between 18 and 65 years
* Both sexes
* Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS > 100)
* Expanded Disability Status Scale (EDSS between 3 and 6 inclusive)
* Berg Balance Scale (BBS ≥ 46)
* Indication for the use of the Exoband orthosis for gait assistance
* Modified Fatigue Impact Scale (MFIS) physical subscale ≤ 20
* Signed informed consent

Exclusion Criteria:

* Presence of severe or current visual or auditory impairments
* Relapses within the last 3 months
* Presence of severe anxiety or depression
* Severe spasticity patterns in the lower limbs or fixed distal tendon contractures
* Presence of motion sickness symptoms induced by virtual reality (VR)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Score of the standardized tests and gait parameters | From T1 (day 2) to T2 (day 9)
  This outcome assesses the adaptation to the walking brace during ambulation. Gait performance across different sessions will be analyzed and compared to observe improvement between T1 and T2. Participant satisfaction with the use of VR will be considered met if individuals can successfully engage with and complete the sessions using the system.

SECONDARY OUTCOMES:
NASA-TLX (NASA Task Load Index) questionnaire score | T1 (day 2); T2 (day 10); T3 (day 70)
  The NASA-TLX questionnaire score (National Aeronautics and Space Administration Task Load Index) measures physical and mental workload using six items related to mental load, physical activity, speed of performance, performance, effort, and frustration. Each item is accompanied by a 12 cm line scale divided into 20 equal intervals, anchored by binary descriptors (e.g., low/high), delimited by 21 vertical markers, and then converted to a scale from 0 to 100 points. To calculate the score for each scale, the number of lines marked by a participant is counted, 1 is subtracted, and the result is multiplied by 5. Weights from 0-5 will be assigned to the 15 subscale comparisons, which will be multiplied by the corresponding subscale score. The total score (from 0 to 100 points) is estimated by summing the weighted scores and dividing by 15.
MSAQ (Motion Sickness Assessment Questionnaire) questionnaire score | T0 (day 1); T1 (day 2); T2 (day 10)
  The MSAQ questionnaire assesses motion sickness. It consists of 16 questions divided into four subcategories: Gastrointestinal (G), Central (C), Peripheral (P), and Sopite-related (S). Responses are scored on a scale from 1 to 9 points. Each subcategory is scored individually, contributing to a total score ranging from 11 to 144 points. The overall motion sickness score is calculated as the percentage of total points scored: (sum of all item points / 144) × 100. Subscale scores are calculated similarly as percentages within each factor: (sum of gastrointestinal items / 36) × 100; (sum of central items / 45) × 100; (sum of peripheral items / 27) × 100; (sum of sopite items / 36) × 100.
IPQ (iGroupPresence Questionnaire) questionnaire score | T1 (day 2); T2 (day 10)
  The IPQ questionnaire assesses the sense of presence (SOP - level of immersion in VR) of a VR user. The IPQ consists of 14 items divided into four subcategories: spatial presence, involvement, perceived realism level, and a "sense of being present." All items are rated on a seven-point scale (0-6), with a higher score indicating greater SOP. The total score is obtained by summing the scores of individual items (from 0 to 84 points).
MusiQoL (Multiple Sclerosis International Quality of Life) questionnaire score | T1 (day 2), T2 (day 10), T3 (day 70)
  The MusiQoL questionnaire assesses health-related quality of life specifically in individuals with multiple sclerosis. It consists of 31 items grouped into nine dimensions: daily activities, psychological well-being, symptoms, social relationships, family relationships, relationship with healthcare professionals, emotional well-being, intimate relationships, and leisure activities. Each item is rated on a five-point Likert scale (from 1 = "never" to 5 = "always"). Scores for each dimension are calculated as the mean of the corresponding items, then transformed into a 0-100 scale, with higher scores indicating better quality of life.
BBS (Berg Balance Scale) questionnaire score | T1 (day 2); T2 (day 10); T3 (day 70)
  The BBS is a clinical assessment tool used to evaluate balance and fall risk in individuals. It consists of 14 functional tasks, each scored on a scale from 0 (unable to perform) to 4 (normal performance), with a maximum total score of 56 points. The items assess the ability to maintain upright standing positions without support (eyes open, closed, feet together, tandem, single-leg stance), perform posture transitions (e.g., sitting to standing, transfers between bed and chair), turn the body, and complete other tasks requiring static and dynamic postural control.
EDSS (Expanded Disability Status Scale) questionnaire score | T0 (day 1)
  The EDSS is an ordinal rating scale used to quantify disability in individuals with multiple sclerosis. Scores range from 0 (normal neurological status) to 10 (death due to MS), with 0.5-point increments indicating increasing levels of disability. The scale evaluates several functional systems, including motor, sensory, visual, bowel and bladder functions, and cognitive impairments, providing an overall measure of disability.
MFIS (Modified Fatigue Impact Scale) questionnaire score | T0 (day 1); T1 (day 2); Th (day 3-9); T2 (day 10); T3 (day 70)
  The MFIS is a 21-item self-report questionnaire that assesses the perceived impact of fatigue on daily life, covering three domains: physical (0-36), cognitive (0-40), and psychosocial (0-8). Each item is rated from 0 to 4. The total score ranges from 0 to 84, with higher scores indicating greater fatigue impact. Subscale scores provide domain-specific insights, useful for monitoring targeted therapeutic interventions.
MSWS-12 (Twelve-Item Multiple Sclerosis Walking Scale) questionnaire score | T1 (day 2); T2 (day 10); T3 (day 70)
  The MSWS-12 is a self-reported questionnaire designed to measure the impact of MS on walking ability. It consists of 12 items rated on a 5-point scale (1-5), reflecting perceived walking difficulties over the past two weeks. Assessed domains include balance, speed, walking distance, and need for assistance. The total raw score is converted to a 0-100 scale, with higher scores indicating greater walking disability.
Timed 25-Foot Walk Test (T25FW) test score | T1 (day 2); T2 (day 10); T3 (day 70)
  The T25FW assesses walking speed and is used to evaluate the walking ability of individuals with multiple sclerosis. The test involves the participant walking 25 feet (approximately 7.62 meters) as quickly as possible, performing two separate trials. The time taken to complete each trial is measured in seconds using a stopwatch. The final score is calculated by averaging the two recorded times.
2MWT (2-Minute Walk Test) test score | T1 (day 2); T2 (day 10); T3 (day 70)
  The 2MWT is a test used to assess walking ability, in which the subject is asked to walk as fast as possible for 2 minutes on a flat surface. The total distance covered during this time is measured. The test evaluates walking speed, as well as the patient's cardiovascular and muscular endurance.
TAM (Technology Acceptance Model) questionnaire score | T0 (day 1); T2 (day 10)
  The TAM is a tool used to measure users' acceptance of technology, based on two key components: perceived usefulness (how much the user believes the technology improves their performance) and perceived ease of use (how easy the user finds the technology to use). The test includes 12 items scored from 1 to 4, with a total score of 48. Higher scores indicate lower acceptance of the technology.
TLSQ-WT (Tele-healthcare Satisfaction Questionnaire - Wearable Technology) questionnaire score | T2 (day 10)
  The TLSQ-WT is an assessment tool designed to measure patients' satisfaction with telemedicine services. It evaluates six dimensions of the user experience with the wearable component of a system: Benefits, Usability, Self-perception, Privacy and Loss of Control, Quality of Life, and Comfort of Use.
  Each area includes five statements rated by the user on a 5-point Likert scale from 0 (strongly disagree) to 4 (strongly agree), for a total of 30 items. The final score ranges from 0 to 120.
Timed Up and Go (TUG) test score | T1 (day 2); T2 (day 10); T3 (day 70)
  The TUG (Podsiadlo & Richardson, 1991) is a functional test commonly used to assess mobility and fall risk in patients with neurological conditions, including multiple sclerosis. The test involves asking the patient to stand up from a chair, walk 3 meters, turn around, walk back, and sit down again. The time required to complete the task is recorded in seconds using a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Loredana Sabattini, Principal Investigator — IRCCS Istituto delle Scienze Neurologiche di Bologna - AUSL of Bologna
Locations (1):
- IRCCS Istituto delle Scienze Neurologiche di Bologna - AUSL of Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsai MF, Bandini A, Wang RH, Zariffa J. Capturing Representative Hand Use at Home Using Egocentric Video in Individuals with Upper Limb Impairment. J Vis Exp. 2020 Dec 23;(166). doi: 10.3791/61898. PMID 33427235
- [Background] Casuso-Holgado MJ, Martin-Valero R, Carazo AF, Medrano-Sanchez EM, Cortes-Vega MD, Montero-Bancalero FJ. Effectiveness of virtual reality training for balance and gait rehabilitation in people with multiple sclerosis: a systematic review and meta-analysis. Clin Rehabil. 2018 Sep;32(9):1220-1234. doi: 10.1177/0269215518768084. Epub 2018 Apr 13. PMID 29651873
- [Background] Peruzzi A, Cereatti A, Della Croce U, Mirelman A. Effects of a virtual reality and treadmill training on gait of subjects with multiple sclerosis: a pilot study. Mult Scler Relat Disord. 2016 Jan;5:91-6. doi: 10.1016/j.msard.2015.11.002. Epub 2015 Nov 6. PMID 26856951
- [Background] Bettoni E, Ferriero G, Bakhsh H, Bravini E, Massazza G, Franchignoni F. A systematic review of questionnaires to assess patient satisfaction with limb orthoses. Prosthet Orthot Int. 2016 Apr;40(2):158-69. doi: 10.1177/0309364614556836. Epub 2014 Nov 26. PMID 25428901
- [Background] Marimon X, Mengual I, Lopez-de-Celis C, Portela A, Rodriguez-Sanz J, Herraez IA, Perez-Bellmunt A. Kinematic Analysis of Human Gait in Healthy Young Adults Using IMU Sensors: Exploring Relevant Machine Learning Features for Clinical Applications. Bioengineering (Basel). 2024 Jan 23;11(2):105. doi: 10.3390/bioengineering11020105. PMID 38391591
- [Background] Panizzolo FA, Cimino S, Pettenello E, Belfiore A, Petrone N, Marcolin G. Effect of a passive hip exoskeleton on walking distance in neurological patients. Assist Technol. 2022 Sep 3;34(5):527-532. doi: 10.1080/10400435.2021.1880494. Epub 2021 Mar 5. PMID 33481693
- [Background] Karunakaran KK, Pamula SD, Bach CP, Legelen E, Saleh S, Nolan KJ. Lower extremity robotic exoskeleton devices for overground ambulation recovery in acquired brain injury-A review. Front Neurorobot. 2023 May 25;17:1014616. doi: 10.3389/fnbot.2023.1014616. eCollection 2023. PMID 37304666
- [Background] Homayuni A, Abedini S, Hosseini Z, Etemadifar M, Ghanbarnejad A. Explaining the facilitators of quality of life in patients with multiple sclerosis: a qualitative study. BMC Neurol. 2021 May 11;21(1):193. doi: 10.1186/s12883-021-02213-9. PMID 33975555
- [Background] Gil-Gonzalez I, Martin-Rodriguez A, Conrad R, Perez-San-Gregorio MA. Quality of life in adults with multiple sclerosis: a systematic review. BMJ Open. 2020 Nov 30;10(11):e041249. doi: 10.1136/bmjopen-2020-041249. PMID 33257490